CLINICAL TRIAL: NCT03035630
Title: Randomized Phase II Trial Comparing Sequential First-line Sunitinib and Second-line Avelumab vs First-line Avelumab and Second-line Sunitinib for Metastatic Renal Cell Carcinoma: SUAVE Trial. Hoosier Cancer Research Network GU15-223
Brief Title: Sunitinib Followed by Avelumab or the Reverse for Metastatic Renal Cell Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal investigator left lead institution and efforts to open the protocol at another institution were not successful.
Sponsor: Guru Sonpavde (Other)
Collaborators: Hoosier Cancer Research Network (Other); Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Guru Sonpavde, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GU15-223
Record Dates: First submitted 2017-01-24; First posted 2017-01-30 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Clear-cell Renal Cell Carcinoma; RCC; Kidney Cancer; Clear-cell Kidney Carcinoma
Keywords: Avelumab; Sunitinib; MSB0010718C; Sutent; IgG1 antibody; Anti-PD-L1; Tyrosine kinase inhibitor
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — avelumab; Sunitinib

STUDY DESIGN:
Masking Description: Open-Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Avelumab then Sunitinib for Investigational Arm A (Experimental): First-Line Medication:
  * Avelumab 10mg/kg IV on D1 and D15 of every 28 day cycle, until irRECIST 1.1 disease progression criteria is documented.
    * Subjects will have a mandatory an inter-line washout period (14-60 days) before receiving first dose of second-line medication.
  Second-Line Medication:
  * Sunitinib 50 mg po once daily from D1 to D14 of every 21 day cycle until RECIST 1.1 disease progression criteria is documented.
  Subjects who do not have disease progression at end of first-line treatment and are removed due to toxicities or personal decision, may switch to either the second-line therapy or be monitored during the inter-line period until progression, which may be longer than 60 days.
  Interventions: Drug: Avelumab; Drug: Sunitinib
- Sunitinib then Avelumab for Investigational Arm B (Experimental): First-Line Medication:
  * Sunitinib 50 mg po once daily from D1 to D14 of every 21 day cycle until RECIST 1.1 disease progression criteria is documented.
    * Subjects will have a mandatory inter-line washout period (14-60 days) before receiving first dose of second-line medication.
  Second-Line Medication:
  * Avelumab 10mg/kg IV on D1 and D15 of every 28 day cycle, until irRECIST 1.1 disease progression criteria is documented.
  Subjects who do not have disease progression at end of first-line treatment and are removed due to toxicities or personal decision, may switch to either the second-line therapy or be monitored during the inter-line period until progression, which may be longer than 60 days.
  Interventions: Drug: Avelumab; Drug: Sunitinib

INTERVENTIONS:
Drug: Avelumab — Avelumab 10mg/kg IV over 60 minutes on D1 and D15 of every 28 day cycle
  Other Names: MSB0010718C
Drug: Sunitinib — Sunitinib 50 mg once daily from D1 to D14 of every 21 day cycle
  Other Names: Sutent

SUMMARY:
This is an open label, randomized phase II trial. Eligible subjects will be randomized in a 1:1 ratio and stratified for known prognostics variables to one of two first-line medication treatment arms. Once disease progression has been documented, and following a required inter-line washout period, subjects will receive either second-line medication treatment or discontinue treatment, per discretion of treating investigator.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center trial. Eligible subjects will be randomized and stratified to one of two arms:

FIRST-LINE INVESTIGATIONAL TREATMENT ARM A:

* Avelumab 10mg/kg intravenously (IV) on Day 1 (D1) and Day 15 (D15) of every 28 day cycle until documented disease progression per Immune-related Response Evaluation Criteria In Solid Tumors (irRECIST) 1.1

SECOND-LINE INVESTIGATIONAL TREATMENT ARM A:

* Following completion of an inter-line washout period of a minimum of 2 weeks up to a maximum of 60 days (or at the discretion of treating investigator) subjects will receive:

  * Sunitinib 50 mg by mouth (po) once daily from D1 to D14 of every 21 day cycle until documented disease progression per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 OR
  * Discontinue treatment

FIRST-LINE INVESTIGATIONAL TREATMENT ARM B:

* Sunitinib 50 mg po once daily from D1 to D14 of every 21 day cycle until documented disease progression per RECIST 1.1

SECOND-LINE INVESTIGATIONAL TREATMENT ARM B:

* Following completion of an inter-line washout period of a minimum of 2 weeks up to a maximum of 60 days (or at the discretion of treating investigator) subjects will receive:

  * Avelumab 10mg/kg IV on D1 and D15 every 28 day cycle until documented disease progression per irRECIST 1.1 OR
  * Discontinue treatment

NOTE:

Subjects who do not experience disease progression at end of first-line treatment and are removed from first-line treatment due to toxicities or personal decision, may also either receive second-line therapy or be monitored during the inter-line period until progression (which may be longer than 60 days) per discretion of treating investigator.

Radiological disease evaluation assessments will be completed every 12 weeks.

To demonstrate adequate organ function, all screening labs must be obtained within 14 days prior to registration:

Hematological:

* Absolute Neutrophil Count (ANC) ≥ 1.5 K/mm3
* Hemoglobin (Hgb) ≥ 9 g/dL
* Platelets ≥ 100 K/ mm3

Renal:

* Calculated creatinine clearance by Cockcroft-Gault formula ≥ 40 ml/min

Hepatic:

* Bilirubin ≤ 1.5 × upper limit of normal (ULN)
* Aspartate aminotransferase (AST) ≤ 2.5 × ULN
* Alanine aminotransferase (ALT) ≤ 2.5 × ULN

Miscellaneous:

* Urine/serum pregnancy test - Negative

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following applicable inclusion criteria to participate in this study:

* Written informed consent and HIPAA authorization for release of personal health information prior to registration.
* Age ≥ 18 years at the time of consent.
* Karnofsky performance status ≥ 60 within 28 days prior to registration.
* Histological or cytological confirmation of ccRCC (component of clear cell histology required).
* Measurable metastatic disease according to RECIST 1.1 criteria within 28 days prior to registration.
* Received no prior mTOR or PD1/PD-L1 inhibitors (prior IL-2 is allowed). Prior VEGF inhibitor is allowed only if >12 months prior to registration, and only if earlier if administered in the neoadjuvant or adjuvant setting
* Females of childbearing potential must have a negative serum pregnancy test within 14 days prior to registration. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months
* Females of childbearing potential and males must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception from the time of informed consent until 60 days after treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study

Exclusion Criteria:

Subjects meeting any of the criteria below may not participate in the study:

* Active infection requiring systemic therapy.
* Known HIV positive (HIV testing is not required for eligibility)
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* Known additional invasive malignancy that is active and/or progressive requiring treatment; exceptions include locally curable cancers, or other cancer for which the subject has been disease-free for at least three years or prostate cancer on surveillance.
* Active central nervous system (CNS) metastases (previously treated CNS metastasis are allowed if subject completed radiation ≥2 weeks earlier and off steroids, and neurologically stable or subject has been on requiring ≤10 mg of daily prednisone or prednisone equivalent dose of another corticosteroid for ≥2 weeks) is acceptable)
* Treatment with any investigational agent (chemotherapy or biologic treatment) within 28 days prior to registration.
* Subjects who have not recovered from toxicities from prior systemic anti-cancer treatment or local therapies (a residual toxicity likely to be chronic but controlled and manageable is allowed, e.g. endocrine syndromes from prior interleukin-2).
* Subjects who have undergone major surgery < 4 weeks or minor surgery < 2 weeks prior to registration. Wounds must be completely healed prior to study entry and subjects must have recovered from all toxicities from surgery. NOTE: placement of a vascular access device is not considered major or minor surgery in this regard.
* Prior radiation therapy is allowed as long as irradiated area was not the sole source of measurable disease and radiotherapy was completed with recovery from toxicity, at least 2 weeks prior to registration, and subject has recovered from toxicity. If the irradiated area is the only site of disease, there must be evidence of progressive disease outside of the radiation field .
* Uncontrolled adrenal insufficiency
* Any active known or suspected autoimmune disease
* Recent or active bleeding diathesis or arterial vascular event (including embolic arterial event such as cerebrovascular accident (or transient ischemic attacks) within 6 months of registration. NOTE: subjects with deep venous thrombosis or pulmonary embolism allowed even within 6 months if controlled on anticoagulation (such as warfarin or heparin provided that their medication dose and INR/PTT are stable)
* Previous assignment to treatment during this study. Subjects permanently withdrawn from study participation will not be allowed to re-enter the study
* Uncontrolled hypertension (systolic pressure > 140 mm Hg or diastolic pressure > 90 mm Hg on repeated measurement) despite optimal medical management.
* Active or clinically significant cardiac disease within 6 months including:

  * Symptomatic Congestive heart failure - New York Heart Association (NYHA)

    > Class II
  * Symptomatic Coronary artery disease (controlled clinically on medication allowed)
  * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin. Controlled atrial fibrillation is allowed.
  * Unstable angina or myocardial infarction.
* Any hemorrhage or bleeding event ≥ NCI CTCAE v4 Grade 3 within 4 weeks prior to start of study medication.
* Subjects with any previously untreated or concurrent cancer that is distinct in primary site or histology from ccRCC except cervical cancer in-situ, treated localized basal cell carcinoma, Gleason score 6 prostate cancer or superficial bladder tumor.
* Known current or chronic hepatitis B or C infection requiring treatment with antiviral therapy. (NOTE: testing not required)
* Presence of non-healing wound, non-healing ulcer or bone fracture.
* Renal failure requiring hemo- or peritoneal dialysis.
* Persistent proteinuria ≥ Grade 3 NCI-CTCAE v4 (> 3.5 g/24hrs, measured by urine protein: creatinine ratio on a random urine sample)
* Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)."
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
* Pleural effusion or ascites that causes respiratory compromise (≥ Grade 2 dyspnea NCI-CTCAE v4)
* History of organ allograft (including corneal transplant)
* Known or suspected allergy or hypersensitivity to any drugs, study drug classes, or excipients of the formulations given during the course of this trial.
* Any uncontrolled malabsorption condition
* Any condition which in the site investigator's opinion, makes the subject unsuitable for trial participation.
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Overall Progression-Free Survival (PFS) | up to 24 months
  Compare PFS1 + PFS2 rates for overall PFS

SECONDARY OUTCOMES:
Overall Failure-Free Survival (FFS) | up to 24 months
  Compare FFS1 rates for first-line therapy on each arm
Overall Survival (OS) | up to 36 months
  Compare OS rates for subjects on each arm
Overall Response Rate (RR) | 2 years
  Compare RR and PFS1 of sunitinib vs. avelumab as first-line therapy and PFS2 as second-line therapy
Overall Toxicities | up to 36 months
  Describe toxicities of sunitinib and avelumab

CONTACTS AND LOCATIONS:
Overall Officials: Guru Sonpavde, M.D., Study Chair — Hoosier Cancer Research Network
Locations (1):
- University of Alabama Hematology Oncology Clinic at Medical West, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Hoosier Cancer Research Network Website — http://www.hoosiercancer.org